CLINICAL TRIAL: NCT05439421
Title: Consumer Perceptions of Waterpipe Tobacco Packaging and Digital Marketing Claims
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00060111; R01CA239192 (NIH)
Record Dates: First submitted 2022-06-22; First posted 2022-06-30 (Actual); Results first posted 2023-11-15 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2023-08

CONDITIONS: Waterpipe Tobacco Smoking
Keywords: Waterpipe tobacco smoking; hookah tobacco warning; hookah tobacco
MeSH Terms: interventions — Drug Packaging

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to see 6 packages and 10 advertisements, with or without the claim of interest on each.
Who Masked: Participant
Masking Description: Participants will be blinded to which stimuli have the claims of interest and which do not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (32):
- With Claim 0% Tar (Experimental): Package or digital marketing advertisement containing claim of interest
  Interventions: Behavioral: Package/Advertisement With Claim
- Without Claim 0% Tar (Experimental): Package or digital marketing advertisement without claim of interest
  Interventions: Behavioral: Package/Advertisement Without Claim
- With Claim No Chemicals (Experimental): Package or digital marketing advertisement containing claim of interest
  Interventions: Behavioral: Package/Advertisement With Claim
- Without Claim No Chemicals (Experimental): Package or digital marketing advertisement without claim of interest
  Interventions: Behavioral: Package/Advertisement Without Claim
- With Claim Apple Image (Experimental): Package or digital marketing advertisement containing claim of interest
  Interventions: Behavioral: Package/Advertisement With Claim
- Without Claim Apple Image (Experimental): Package or digital marketing advertisement without claim of interest
  Interventions: Behavioral: Package/Advertisement Without Claim
- With Claim 100% Food Grade Glycerin (Experimental): Package or digital marketing advertisement containing claim of interest
  Interventions: Behavioral: Package/Advertisement With Claim
- Without Claim 100% Food Grade Glycerin (Experimental): Package or digital marketing advertisement without claim of interest
  Interventions: Behavioral: Package/Advertisement Without Claim
- With Claim Ultra Light (Experimental): Package or digital marketing advertisement containing claim of interest
  Interventions: Behavioral: Package/Advertisement With Claim
- Without Claim Ultra Light (Experimental): Package or digital marketing advertisement without claim of interest
  Interventions: Behavioral: Package/Advertisement Without Claim
- With Claim Fresh Hookah Tobacco (Experimental): Package or digital marketing advertisement containing claim of interest
  Interventions: Behavioral: Package/Advertisement With Claim
- Without Claim Fresh Hookah Tobacco (Experimental): Package or digital marketing advertisement without claim of interest
  Interventions: Behavioral: Package/Advertisement Without Claim
- With Claim Lower Nicotine Tobacco (Experimental): Package or digital marketing advertisement containing claim of interest
  Interventions: Behavioral: Package/Advertisement With Claim
- Without Claim Lower Nicotine Tobacco (Experimental): Package or digital marketing advertisement without claim of interest
  Interventions: Behavioral: Package/Advertisement Without Claim
- With Claim Premium Shisha Tobacco (Experimental): Package or digital marketing advertisement containing claim of interest
  Interventions: Behavioral: Package/Advertisement With Claim
- Without Claim Premium Shisha Tobacco (Experimental): Package or digital marketing advertisement without claim of interest
  Interventions: Behavioral: Package/Advertisement Without Claim
- With Claim High Quality Shisha Tobacco (Experimental): Package or digital marketing advertisement containing claim of interest
  Interventions: Behavioral: Package/Advertisement With Claim
- Without Claim High Quality Shisha Tobacco (Experimental): Package or digital marketing advertisement without claim of interest
  Interventions: Behavioral: Package/Advertisement Without Claim
- With Claim Don't blow smoke - blow clouds (Experimental): Package or digital marketing advertisement containing claim of interest
  Interventions: Behavioral: Package/Advertisement With Claim
- Without Claim Don't blow smoke - blow clouds (Experimental): Package or digital marketing advertisement without claim of interest
  Interventions: Behavioral: Package/Advertisement Without Claim
- With Claim Contains natural, unwashed tobacco leaf (Experimental): Package or digital marketing advertisement containing claim of interest
  Interventions: Behavioral: Package/Advertisement With Claim
- Without Claim Contains natural, unwashed tobacco leaf (Experimental): Package or digital marketing advertisement without claim of interest
  Interventions: Behavioral: Package/Advertisement Without Claim
- With Claim We only use ingredients which are FDA approved (Experimental): Package or digital marketing advertisement containing claim of interest
  Interventions: Behavioral: Package/Advertisement With Claim
- Without Claim We only use ingredients which are FDA approved (Experimental): Package or digital marketing advertisement without claim of interest
  Interventions: Behavioral: Package/Advertisement Without Claim
- With Claim Passing flavored tobacco smoke through water cools and purifies it (Experimental): Package or digital marketing advertisement containing claim of interest
  Interventions: Behavioral: Package/Advertisement With Claim
- Without Claim Passing flavored tobacco smoke through water cools and purifies it (Experimental): Package or digital marketing advertisement without claim of interest
  Interventions: Behavioral: Package/Advertisement Without Claim
- With Claim Natural flavor (Experimental): Package or digital marketing advertisement containing claim of interest
  Interventions: Behavioral: Package/Advertisement With Claim
- Without Claim Natural flavor (Experimental): Package or digital marketing advertisement without claim of interest
  Interventions: Behavioral: Package/Advertisement Without Claim
- With Claim Shisha or hookah tobacco is unique and completely unlike that found in cigarettes (Experimental): Package or digital marketing advertisement containing claim of interest
  Interventions: Behavioral: Package/Advertisement With Claim
- Without Claim Shisha or hookah tobacco is unique and completely unlike that found in cigarettes (Experimental): Package or digital marketing advertisement without claim of interest
  Interventions: Behavioral: Package/Advertisement Without Claim
- With Claim water in the shisha effectively cools and filters the smoke, making smooth and light (Experimental): Package or digital marketing advertisement containing claim of interest
  Interventions: Behavioral: Package/Advertisement With Claim
- Without Claim water in the shisha effectively cools and filters the smoke, making smooth and light (Experimental): Package or digital marketing advertisement without claim of interest
  Interventions: Behavioral: Package/Advertisement Without Claim

INTERVENTIONS:
Behavioral: Package/Advertisement With Claim — Waterpipe tobacco packages and digital marketing advertisement images with claim of interest as part of design
  Arms: With Claim 0% Tar; With Claim 100% Food Grade Glycerin; With Claim Apple Image; With Claim Contains natural, unwashed tobacco leaf; With Claim Don't blow smoke - blow clouds; With Claim Fresh Hookah Tobacco; With Claim High Quality Shisha Tobacco; With Claim Lower Nicotine Tobacco; With Claim Natural flavor; With Claim No Chemicals; With Claim Passing flavored tobacco smoke through water cools and purifies it; With Claim Premium Shisha Tobacco; With Claim Shisha or hookah tobacco is unique and completely unlike that found in cigarettes; With Claim Ultra Light; With Claim We only use ingredients which are FDA approved; With Claim water in the shisha effectively cools and filters the smoke, making smooth and light
Behavioral: Package/Advertisement Without Claim — Waterpipe tobacco packages and digital marketing advertisements shown without claim of interest as part of design
  Arms: Without Claim 0% Tar; Without Claim 100% Food Grade Glycerin; Without Claim Apple Image; Without Claim Contains natural, unwashed tobacco leaf; Without Claim Don't blow smoke - blow clouds; Without Claim Fresh Hookah Tobacco; Without Claim High Quality Shisha Tobacco; Without Claim Lower Nicotine Tobacco; Without Claim Natural flavor; Without Claim No Chemicals; Without Claim Passing flavored tobacco smoke through water cools and purifies it; Without Claim Premium Shisha Tobacco; Without Claim Shisha or hookah tobacco is unique and completely unlike that found in cigarettes; Without Claim Ultra Light; Without Claim We only use ingredients which are FDA approved; Without Claim water in the shisha effectively cools and filters the smoke, making smooth and light

SUMMARY:
The purpose of the study is to evaluate the impact of marketing claims commonly found on waterpipe, also known as hookah, tobacco packages and in digital marketing on young adults' willingness to try hookah tobacco. Participants will complete two tasks, in random order. Participants will view six sample waterpipe tobacco packages, randomized at the package level to contain a prohibited or potentially-prohibited claim or not (Packaging Task). In the other task, they will view 10 digital marketing advertisements (i.e. Instagram posts or website pages) either with or without prohibited or potentially-prohibited claim, randomized at the advertisements level (Digital Marketing Task).

DETAILED DESCRIPTION:
Background/Objectives The Food and Drug Administration (FDA) has begun to prohibit certain claims on Waterpipe Tobacco (WT) packaging and advertising. Under Section 911 of the Family Smoking Prevention and Tobacco Control Act, manufacturers and retailers are prohibited from making unauthorized modified risk tobacco product (MRTP) claims, including statements that the product or its smoke: (1) results in reduced harm; (2) contains a reduced level of a substance or presents a reduced exposure to a substance; (3) does not contain or is free of a substance; and (4) statements that use modified risk descriptors such as light, mild, low, or similar descriptors. Some prohibited claims are easily identifiable, but others are more difficult to identify due to lack of specificity in the law and the implicit nature of some claims. Evidence is needed specific to WT packaging and marketing to determine which claims may be associated with consumer harm misperceptions to inform future regulatory actions. The study will address this gap by assessing how such claims influence consumer perceptions and behavioral intentions.

ELIGIBILITY:
Inclusion Criteria:

* United States (U.S.) Resident
* Has used waterpipe tobacco within the past year (self-report)
* Has not used waterpipe tobacco within the past year but it susceptible to use (self- report)

Exclusion Criteria:

* Younger than 18 or older than 29
* Non U.S. Resident
* Has not used waterpipe tobacco within in the past year and is not susceptible to use (self-report)

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1507 (Actual)
Dates: Start 2022-10-25 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2022-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin Sutfin, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized to see 6 packages and 10 advertisements with/without the claim of interest on each (32 arms). The randomization was repeated prior to each claim of interest. 1507 unique were enrolled in total.
Groups:
- With Claim: Package or digital marketing advertisement containing claim of interest Package/Advertisement With Claim: Waterpipe tobacco packages and digital marketing advertisement images with claim of interest as part of design
- Without Claim: Package or digital marketing advertisement without claim of interest Package/Advertisement Without Claim: Waterpipe tobacco packages and digital marketing advertisements shown without claim of interest as part of design
Period: Zero Percent Tar
Arm/Group | With Claim | Without Claim
Started | 742 | 765
Completed | 742 | 765
Not Completed | 0 | 0
Period: No Chemicals
Arm/Group | With Claim | Without Claim
Started | 764 | 743
Completed | 764 | 743
Not Completed | 0 | 0
Period: Apple Image
Arm/Group | With Claim | Without Claim
Started | 743 | 764
Completed | 743 | 764
Not Completed | 0 | 0
Period: Hundred Percent Food Grade Glycerin
Arm/Group | With Claim | Without Claim
Started | 746 | 761
Completed | 746 | 761
Not Completed | 0 | 0
Period: Ultra Light
Arm/Group | With Claim | Without Claim
Started | 731 | 776
Completed | 731 | 776
Not Completed | 0 | 0
Period: Fresh Hookah Tobacco
Arm/Group | With Claim | Without Claim
Started | 706 | 801
Completed | 706 | 801
Not Completed | 0 | 0
Period: Lower Nicotine Tobacco
Arm/Group | With Claim | Without Claim
Started | 742 | 765
Completed | 742 | 765
Not Completed | 0 | 0
Period: Premium Shisha Tobacco
Arm/Group | With Claim | Without Claim
Started | 764 | 743
Completed | 764 | 743
Not Completed | 0 | 0
Period: High Quality Shisha Tobacco
Arm/Group | With Claim | Without Claim
Started | 743 | 764
Completed | 743 | 764
Not Completed | 0 | 0
Period: Don't Blow Smoke - Blow Clouds
Arm/Group | With Claim | Without Claim
Started | 746 | 761
Completed | 746 | 761
Not Completed | 0 | 0
Period: Contains Natural, Unwashed Tobacco Leaf
Arm/Group | With Claim | Without Claim
Started | 731 | 776
Completed | 731 | 776
Not Completed | 0 | 0
Period: We Only Use FDA Approved Ingredients
Arm/Group | With Claim | Without Claim
Started | 706 | 801
Completed | 706 | 801
Not Completed | 0 | 0
Period: H2O Cools Puirfies Tobacco Smoke
Arm/Group | With Claim | Without Claim
Started | 753 | 754
Completed | 753 | 754
Not Completed | 0 | 0
Period: Natural Flavor
Arm/Group | With Claim | Without Claim
Started | 783 | 724
Completed | 783 | 724
Not Completed | 0 | 0
Period: Shisha/Hookah Tobacco is Unique
Arm/Group | With Claim | Without Claim
Started | 749 | 758
Completed | 749 | 758
Not Completed | 0 | 0
Period: Shisha H2O Cools and Filters Smoke
Arm/Group | With Claim | Without Claim
Started | 722 | 785
Completed | 722 | 785
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants were randomized to see 6 packages and 10 advertisements with/without the claim of interest on each (32 arms). The randomization was repeated prior to each claim of interest. 1507 unique were enrolled in total.
Groups:
- With Claim: Package or digital marketing advertisement containing claim of interest Package / Advertisement With Claim: Waterpipe tobacco packages and digital marketing advertisement images with claim of interest as part of design
- Without Claim: Package or digital marketing advertisement without claim of interest Package / Advertisement Without Claim: Waterpipe tobacco packages and digital marketing advertisements shown without claim of interest as part of design
- Total: Total of all reporting groups
Arm/Group | With Claim | Without Claim | Total
Number analyzed (Participants) | 742 | 765 | 1507
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.1 (3.2) | 24.7 (3.2) | 24.9 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 481 | 488 | 969
  Male | 261 | 277 | 538
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 167 | 163 | 330
  Not Hispanic or Latino | 575 | 602 | 1177
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 9 | 15
  Asian | 56 | 60 | 116
  Native Hawaiian or Other Pacific Islander | 4 | 2 | 6
  Black or African American | 163 | 182 | 345
  White | 432 | 429 | 861
  More than one race | 31 | 32 | 63
  Unknown or Not Reported | 50 | 51 | 101

OUTCOME MEASURES:

1. Primary Outcome: Willingness to Try Hookah Tobacco (Packaging Task )
Description: One item to assess the extent to which young adults are willing to try the waterpipe tobacco product: How likely would you be to try this specific product?
  Response scale: (1) Not at all likely to (4) Very likely
Time Frame: minute 5
Population: Only certain Arms involved the Packaging Experiment
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | With Claim 0% Tar | Without Claim 0% Tar | With Claim No Chemicals | Without Claim No Chemicals | With Claim Apple Image | Without Claim Apple Image | With Claim 100% Food Grade Glycerin | Without Claim 100% Food Grade Glycerin | With Claim Ultra Light | Without Claim Ultra Light | With Claim Fresh Hookah Tobacco | Without Claim Fresh Hookah Tobacco | With Claim Lower Nicotine Tobacco | Without Claim Lower Nicotine Tobacco | With Claim Premium Shisha Tobacco | Without Claim Premium Shisha Tobacco | With Claim High Quality Shisha Tobacco | Without Claim High Quality Shisha Tobacco | With Claim Don't Blow Smoke - Blow Clouds | Without Claim Don't Blow Smoke - Blow Clouds | With Claim Contains Natural, Unwashed Tobacco Leaf | Without Claim Contains Natural, Unwashed Tobacco Leaf | With Claim We Only Use Ingredients Which Are FDA Approved | Without Claim We Only Use Ingredients Which Are FDA Approved | With Claim Passing Flavored Tobacco Smoke Through Water Cools and Purifies it | Without Claim Passing Flavored Tobacco Smoke Through Water Cools and Purifies it | With Claim Natural Flavor | Without Claim Natural Flavor | With Claim Shisha or Hookah Tobacco is Unique and Completely Unlike That Found in Cigarettes | Without Claim Shisha or Hookah Tobacco is Unique and Completely Unlike That Found in Cigarettes | With Claim Water in the Shisha Effectively Cools and Filters the Smoke, Making Smooth and Light | Without Claim Water in the Shisha Effectively Cools and Filters the Smoke, Making Smooth and Light
Number analyzed (Participants) | 742 | 765 | 764 | 743 | 743 | 764 | 746 | 761 | 731 | 776 | 706 | 801 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
score on a scale | 1.9 (0.05) | 1.87 (0.05) | 1.9 (0.06) | 1.63 (0.05) | 1.95 (0.06) | 1.78 (0.05) | 1.81 (0.05) | 1.79 (0.05) | 1.84 (0.06) | 1.81 (0.05) | 1.86 (0.06) | 1.80 (0.05) |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |

2. Primary Outcome: Willingness to Smoke Hookah Tobacco (Digital Marketing Task )
Description: One item to assess the extent to which young adults want to try smoking hookah: How much does this advertisement make you want to smoke hookah?
  Response scale: (1) Not at all to (4) A lot
Time Frame: minute 5
Population: Only certain Arms involved the Digital Marketing Experiment
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | With Claim 0% Tar | Without Claim 0% Tar | With Claim No Chemicals | Without Claim No Chemicals | With Claim Apple Image | Without Claim Apple Image | With Claim 100% Food Grade Glycerin | Without Claim 100% Food Grade Glycerin | With Claim Ultra Light | Without Claim Ultra Light | With Claim Fresh Hookah Tobacco | Without Claim Fresh Hookah Tobacco | With Claim Lower Nicotine Tobacco | Without Claim Lower Nicotine Tobacco | With Claim Premium Shisha Tobacco | Without Claim Premium Shisha Tobacco | With Claim High Quality Shisha Tobacco | Without Claim High Quality Shisha Tobacco | With Claim Don't Blow Smoke - Blow Clouds | Without Claim Don't Blow Smoke - Blow Clouds | With Claim Contains Natural, Unwashed Tobacco Leaf | Without Claim Contains Natural, Unwashed Tobacco Leaf | With Claim We Only Use Ingredients Which Are FDA Approved | Without Claim We Only Use Ingredients Which Are FDA Approved | With Claim Passing Flavored Tobacco Smoke Through Water Cools and Purifies it | Without Claim Passing Flavored Tobacco Smoke Through Water Cools and Purifies it | With Claim Natural Flavor | Without Claim Natural Flavor | With Claim Shisha or Hookah Tobacco is Unique and Completely Unlike That Found in Cigarettes | Without Claim Shisha or Hookah Tobacco is Unique and Completely Unlike That Found in Cigarettes | With Claim Water in the Shisha Effectively Cools and Filters the Smoke, Making Smooth and Light | Without Claim Water in the Shisha Effectively Cools and Filters the Smoke, Making Smooth and Light
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 742 | 765 | 764 | 743 | 743 | 764 | 746 | 761 | 731 | 776 | 706 | 801 | 753 | 754 | 783 | 724 | 749 | 758 | 722 | 785
score on a scale |  |  |  |  |  |  |  |  |  |  |  |  | 1.74 (.05) | 1.78 (.05) | 1.46 (.05) | 1.42 (.04) | 1.67 (.05) | 1.75 (.04) | 1.81 (.05) | 1.88 (.05) | 1.74 (.05) | 1.62 (.05) | 1.76 (.05) | 1.69 (.05) | 1.66 (.05) | 1.63 (.05) | 2.00 (.05) | 1.91 (.05) | 1.93 (.05) | 1.78 (.05) | 1.83 (.05) | 1.73 (.05)

3. Other Pre Specified Outcome: Absolute Harm Perception (Packaging Task )
Description: One item to assess young adults' perceptions of how the packaging influences their opinions on the harmfulness of the hookah tobacco: How much does this packaging make you think this product is harmful?
  Response scale: (1) Not at all to (4) A lot
Time Frame: minute 5
Population: Only certain Arms involved the Packaging Experiment
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | With Claim 0% Tar | Without Claim 0% Tar | With Claim No Chemicals | Without Claim No Chemicals | With Claim Apple Image | Without Claim Apple Image | With Claim 100% Food Grade Glycerin | Without Claim 100% Food Grade Glycerin | With Claim Ultra Light | Without Claim Ultra Light | With Claim Fresh Hookah Tobacco | Without Claim Fresh Hookah Tobacco | With Claim Lower Nicotine Tobacco | Without Claim Lower Nicotine Tobacco | With Claim Premium Shisha Tobacco | Without Claim Premium Shisha Tobacco | With Claim High Quality Shisha Tobacco | Without Claim High Quality Shisha Tobacco | With Claim Don't Blow Smoke - Blow Clouds | Without Claim Don't Blow Smoke - Blow Clouds | With Claim Contains Natural, Unwashed Tobacco Leaf | Without Claim Contains Natural, Unwashed Tobacco Leaf | With Claim We Only Use Ingredients Which Are FDA Approved | Without Claim We Only Use Ingredients Which Are FDA Approved | With Claim Passing Flavored Tobacco Smoke Through Water Cools and Purifies it | Without Claim Passing Flavored Tobacco Smoke Through Water Cools and Purifies it | With Claim Natural Flavor | Without Claim Natural Flavor | With Claim Shisha or Hookah Tobacco is Unique and Completely Unlike That Found in Cigarettes | Without Claim Shisha or Hookah Tobacco is Unique and Completely Unlike That Found in Cigarettes | With Claim Water in the Shisha Effectively Cools and Filters the Smoke, Making Smooth and Light | Without Claim Water in the Shisha Effectively Cools and Filters the Smoke, Making Smooth and Light
Number analyzed (Participants) | 742 | 765 | 764 | 743 | 743 | 764 | 746 | 761 | 731 | 776 | 706 | 801 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
score on a scale | 1.74 (0.04) | 1.74 (0.05) | 1.78 (0.05) | 1.67 (0.05) | 1.79 (0.05) | 1.77 (0.05) | 1.82 (0.06) | 1.79 (0.05) | 1.76 (0.05) | 1.72 (0.05) | 1.83 (0.05) | 1.80 (0.05) |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |

4. Other Pre Specified Outcome: Absolute Harm Perception (Digital Marketing Task )
Description: One item to assess young adults' perception of how the advertisement influences their opinions on the harmfulness of smoking hookah: How much does this advertisement make you think smoking hookah is harmful?
  Response scale: (1) Not at all to (4) A lot
Time Frame: minute 5
Population: Only certain Arms involved the Digital Marketing Experiment
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | With Claim 0% Tar | Without Claim 0% Tar | With Claim No Chemicals | Without Claim No Chemicals | With Claim Apple Image | Without Claim Apple Image | With Claim 100% Food Grade Glycerin | Without Claim 100% Food Grade Glycerin | With Claim Ultra Light | Without Claim Ultra Light | With Claim Fresh Hookah Tobacco | Without Claim Fresh Hookah Tobacco | With Claim Lower Nicotine Tobacco | Without Claim Lower Nicotine Tobacco | With Claim Premium Shisha Tobacco | Without Claim Premium Shisha Tobacco | With Claim High Quality Shisha Tobacco | Without Claim High Quality Shisha Tobacco | With Claim Don't Blow Smoke - Blow Clouds | Without Claim Don't Blow Smoke - Blow Clouds | With Claim Contains Natural, Unwashed Tobacco Leaf | Without Claim Contains Natural, Unwashed Tobacco Leaf | With Claim We Only Use Ingredients Which Are FDA Approved | Without Claim We Only Use Ingredients Which Are FDA Approved | With Claim Passing Flavored Tobacco Smoke Through Water Cools and Purifies it | Without Claim Passing Flavored Tobacco Smoke Through Water Cools and Purifies it | With Claim Natural Flavor | Without Claim Natural Flavor | With Claim Shisha or Hookah Tobacco is Unique and Completely Unlike That Found in Cigarettes | Without Claim Shisha or Hookah Tobacco is Unique and Completely Unlike That Found in Cigarettes | With Claim Water in the Shisha Effectively Cools and Filters the Smoke, Making Smooth and Light | Without Claim Water in the Shisha Effectively Cools and Filters the Smoke, Making Smooth and Light
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 742 | 765 | 764 | 743 | 743 | 764 | 746 | 761 | 731 | 776 | 706 | 801 | 753 | 754 | 783 | 724 | 749 | 758 | 722 | 785
score on a scale |  |  |  |  |  |  |  |  |  |  |  |  | 1.90 (.05) | 1.79 (.05) | 1.63 (.05) | 1.67 (.05) | 1.73 (.06) | 1.58 (.04) | 1.86 (.05) | 1.81 (.05) | 1.70 (.05) | 1.61 (.05) | 1.79 (.05) | 1.73 (.05) | 1.80 (.06) | 1.70 (.05) | 1.77 (.05) | 1.59 (.05) | 1.72 (.05) | 1.58 (.04) | 1.71 (.04) | 1.74 (.05)

5. Other Pre Specified Outcome: Product Appeal (Packaging Task )
Description: One item to assess the pictured product's appeal: How appealing is this specific product to you?
  Response scale: (1) Not at all appealing to (4) Very appealing
Time Frame: minute 5
Population: Only certain Arms involved the Packaging Experiment
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | With Claim 0% Tar | Without Claim 0% Tar | With Claim No Chemicals | Without Claim No Chemicals | With Claim Apple Image | Without Claim Apple Image | With Claim 100% Food Grade Glycerin | Without Claim 100% Food Grade Glycerin | With Claim Ultra Light | Without Claim Ultra Light | With Claim Fresh Hookah Tobacco | Without Claim Fresh Hookah Tobacco | With Claim Lower Nicotine Tobacco | Without Claim Lower Nicotine Tobacco | With Claim Premium Shisha Tobacco | Without Claim Premium Shisha Tobacco | With Claim High Quality Shisha Tobacco | Without Claim High Quality Shisha Tobacco | With Claim Don't Blow Smoke - Blow Clouds | Without Claim Don't Blow Smoke - Blow Clouds | With Claim Contains Natural, Unwashed Tobacco Leaf | Without Claim Contains Natural, Unwashed Tobacco Leaf | With Claim We Only Use Ingredients Which Are FDA Approved | Without Claim We Only Use Ingredients Which Are FDA Approved | With Claim Passing Flavored Tobacco Smoke Through Water Cools and Purifies it | Without Claim Passing Flavored Tobacco Smoke Through Water Cools and Purifies it | With Claim Natural Flavor | Without Claim Natural Flavor | With Claim Shisha or Hookah Tobacco is Unique and Completely Unlike That Found in Cigarettes | Without Claim Shisha or Hookah Tobacco is Unique and Completely Unlike That Found in Cigarettes | With Claim Water in the Shisha Effectively Cools and Filters the Smoke, Making Smooth and Light | Without Claim Water in the Shisha Effectively Cools and Filters the Smoke, Making Smooth and Light
Number analyzed (Participants) | 742 | 765 | 764 | 743 | 743 | 764 | 746 | 761 | 731 | 776 | 706 | 801 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
score on a scale | 1.99 (0.05) | 2.01 (0.06) | 1.91 (0.05) | 1.70 (0.05) | 2.01 (0.06) | 1.81 (0.05) | 1.89 (0.05) | 1.84 (0.05) | 1.91 (0.06) | 1.95 (0.05) | 2.02 (0.06) | 1.89 (0.05) |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |

6. Other Pre Specified Outcome: Product Appeal (Digital Marketing Task )
Description: One item to assess the appeal of smoking hookah in the context of the advertisement: How appealing does this advertisement make smoking hookah seem to you?
  Response scale: (1) Not at all appealing to (4) Very appealing
Time Frame: minute 5
Population: Only certain Arms involved the Digital Marketing Experiment
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | With Claim 0% Tar | Without Claim 0% Tar | With Claim No Chemicals | Without Claim No Chemicals | With Claim Apple Image | Without Claim Apple Image | With Claim 100% Food Grade Glycerin | Without Claim 100% Food Grade Glycerin | With Claim Ultra Light | Without Claim Ultra Light | With Claim Fresh Hookah Tobacco | Without Claim Fresh Hookah Tobacco | With Claim Lower Nicotine Tobacco | Without Claim Lower Nicotine Tobacco | With Claim Premium Shisha Tobacco | Without Claim Premium Shisha Tobacco | With Claim High Quality Shisha Tobacco | Without Claim High Quality Shisha Tobacco | With Claim Don't Blow Smoke - Blow Clouds | Without Claim Don't Blow Smoke - Blow Clouds | With Claim Contains Natural, Unwashed Tobacco Leaf | Without Claim Contains Natural, Unwashed Tobacco Leaf | With Claim We Only Use Ingredients Which Are FDA Approved | Without Claim We Only Use Ingredients Which Are FDA Approved | With Claim Passing Flavored Tobacco Smoke Through Water Cools and Purifies it | Without Claim Passing Flavored Tobacco Smoke Through Water Cools and Purifies it | With Claim Natural Flavor | Without Claim Natural Flavor | With Claim Shisha or Hookah Tobacco is Unique and Completely Unlike That Found in Cigarettes | Without Claim Shisha or Hookah Tobacco is Unique and Completely Unlike That Found in Cigarettes | With Claim Water in the Shisha Effectively Cools and Filters the Smoke, Making Smooth and Light | Without Claim Water in the Shisha Effectively Cools and Filters the Smoke, Making Smooth and Light
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 742 | 765 | 764 | 743 | 743 | 764 | 746 | 761 | 731 | 776 | 706 | 801 | 753 | 754 | 783 | 724 | 749 | 758 | 722 | 785
score on a scale |  |  |  |  |  |  |  |  |  |  |  |  | 1.88 (.05) | 1.88 (.05) | 1.53 (.04) | 1.51 (.05) | 1.81 (.05) | 1.89 (.05) | 1.9 (.05) | 2.00 (.06) | 1.86 (.05) | 1.77 (.05) | 1.83 (.05) | 1.78 (.05) | 1.71 (.05) | 1.78 (.05) | 2.09 (.05) | 2.08 (.06) | 2.03 (.05) | 1.93 (.06) | 1.97 (.05) | 1.80 (.05)

7. Other Pre Specified Outcome: Absolute Safety Perception (Packaging Task)
Description: One item to assess young adults' perceptions of how the packaging influences their opinions of how safe the product is: How much does this packaging make you think this product is safe?
  Response scale: (1) Not at all to (4) A lot
Time Frame: minute 5
Population: Only certain Arms involved the Packaging Experiment
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | With Claim 0% Tar | Without Claim 0% Tar | With Claim No Chemicals | Without Claim No Chemicals | With Claim Apple Image | Without Claim Apple Image | With Claim 100% Food Grade Glycerin | Without Claim 100% Food Grade Glycerin | With Claim Ultra Light | Without Claim Ultra Light | With Claim Fresh Hookah Tobacco | Without Claim Fresh Hookah Tobacco | With Claim Lower Nicotine Tobacco | Without Claim Lower Nicotine Tobacco | With Claim Premium Shisha Tobacco | Without Claim Premium Shisha Tobacco | With Claim High Quality Shisha Tobacco | Without Claim High Quality Shisha Tobacco | With Claim Don't Blow Smoke - Blow Clouds | Without Claim Don't Blow Smoke - Blow Clouds | With Claim Contains Natural, Unwashed Tobacco Leaf | Without Claim Contains Natural, Unwashed Tobacco Leaf | With Claim We Only Use Ingredients Which Are FDA Approved | Without Claim We Only Use Ingredients Which Are FDA Approved | With Claim Passing Flavored Tobacco Smoke Through Water Cools and Purifies it | Without Claim Passing Flavored Tobacco Smoke Through Water Cools and Purifies it | With Claim Natural Flavor | Without Claim Natural Flavor | With Claim Shisha or Hookah Tobacco is Unique and Completely Unlike That Found in Cigarettes | Without Claim Shisha or Hookah Tobacco is Unique and Completely Unlike That Found in Cigarettes | With Claim Water in the Shisha Effectively Cools and Filters the Smoke, Making Smooth and Light | Without Claim Water in the Shisha Effectively Cools and Filters the Smoke, Making Smooth and Light
Number analyzed (Participants) | 742 | 765 | 764 | 743 | 743 | 764 | 746 | 761 | 731 | 776 | 706 | 801 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
score on a scale | 1.95 (0.05) | 1.86 (0.05) | 1.89 (0.05) | 1.81 (0.05) | 1.89 (0.05) | 1.80 (0.05) | 1.82 (0.05) | 1.86 (0.05) | 1.89 (0.05) | 1.77 (0.05) | 1.8 (0.05) | 1.8 (0.05) |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |

8. Other Pre Specified Outcome: Absolute Safety Perception (Digital Marketing Task)
Description: One item to assess young adults' perception of how the advertisement influences their opinions on the safety of smoking hookah: How much does this advertisement make you think smoking hookah is safe?
  Response scale: (1) Not at all to (4) A lot
Time Frame: minute 5
Population: Only certain Arms involved the Digital Marketing Experiment
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | With Claim 0% Tar | Without Claim 0% Tar | With Claim No Chemicals | Without Claim No Chemicals | With Claim Apple Image | Without Claim Apple Image | With Claim 100% Food Grade Glycerin | Without Claim 100% Food Grade Glycerin | With Claim Ultra Light | Without Claim Ultra Light | With Claim Fresh Hookah Tobacco | Without Claim Fresh Hookah Tobacco | With Claim Lower Nicotine Tobacco | Without Claim Lower Nicotine Tobacco | With Claim Premium Shisha Tobacco | Without Claim Premium Shisha Tobacco | With Claim High Quality Shisha Tobacco | Without Claim High Quality Shisha Tobacco | With Claim Don't Blow Smoke - Blow Clouds | Without Claim Don't Blow Smoke - Blow Clouds | With Claim Contains Natural, Unwashed Tobacco Leaf | Without Claim Contains Natural, Unwashed Tobacco Leaf | With Claim We Only Use Ingredients Which Are FDA Approved | Without Claim We Only Use Ingredients Which Are FDA Approved | With Claim Passing Flavored Tobacco Smoke Through Water Cools and Purifies it | Without Claim Passing Flavored Tobacco Smoke Through Water Cools and Purifies it | With Claim Natural Flavor | Without Claim Natural Flavor | With Claim Shisha or Hookah Tobacco is Unique and Completely Unlike That Found in Cigarettes | Without Claim Shisha or Hookah Tobacco is Unique and Completely Unlike That Found in Cigarettes | With Claim Water in the Shisha Effectively Cools and Filters the Smoke, Making Smooth and Light | Without Claim Water in the Shisha Effectively Cools and Filters the Smoke, Making Smooth and Light
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 742 | 765 | 764 | 743 | 743 | 764 | 746 | 761 | 731 | 776 | 706 | 801 | 753 | 754 | 4783 | 724 | 749 | 758 | 722 | 785
score on a scale |  |  |  |  |  |  |  |  |  |  |  |  | 1.99 (.05) | 1.69 (.05) | 1.57 (.05) | 1.60 (.04) | 1.73 (.05) | 1.80 (.05) | 1.70 (.05) | 1.67 (.05) | 1.85 (.05) | 1.78 (.05) | 2.10 (.05) | 1.64 (.05) | 1.90 (.05) | 1.72 (.05) | 1.94 (.05) | 1.87 (.06) | 2.15 (.05) | 1.88 (.05) | 1.97 (.06) | 1.88 (.05)

9. Other Pre Specified Outcome: Relative Safety Perception (Packaging Task
Description: One item to assess young adults' perceptions of how safe the product is as compared to other hookah tobacco that might be available to them: Compared to other hookah tobacco on the market, how safe do you think this specific product is? Response scale: (1) Much less safe to (5) Much more safe
Time Frame: minute 5
Population: Only certain Arms involved the Packaging Experiment
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | With Claim 0% Tar | Without Claim 0% Tar | With Claim No Chemicals | Without Claim No Chemicals | With Claim Apple Image | Without Claim Apple Image | With Claim 100% Food Grade Glycerin | Without Claim 100% Food Grade Glycerin | With Claim Ultra Light | Without Claim Ultra Light | With Claim Fresh Hookah Tobacco | Without Claim Fresh Hookah Tobacco | With Claim Lower Nicotine Tobacco | Without Claim Lower Nicotine Tobacco | With Claim Premium Shisha Tobacco | Without Claim Premium Shisha Tobacco | With Claim High Quality Shisha Tobacco | Without Claim High Quality Shisha Tobacco | With Claim Don't Blow Smoke - Blow Clouds | Without Claim Don't Blow Smoke - Blow Clouds | With Claim Contains Natural, Unwashed Tobacco Leaf | Without Claim Contains Natural, Unwashed Tobacco Leaf | With Claim We Only Use Ingredients Which Are FDA Approved | Without Claim We Only Use Ingredients Which Are FDA Approved | With Claim Passing Flavored Tobacco Smoke Through Water Cools and Purifies it | Without Claim Passing Flavored Tobacco Smoke Through Water Cools and Purifies it | With Claim Natural Flavor | Without Claim Natural Flavor | With Claim Shisha or Hookah Tobacco is Unique and Completely Unlike That Found in Cigarettes | Without Claim Shisha or Hookah Tobacco is Unique and Completely Unlike That Found in Cigarettes | With Claim Water in the Shisha Effectively Cools and Filters the Smoke, Making Smooth and Light | Without Claim Water in the Shisha Effectively Cools and Filters the Smoke, Making Smooth and Light
Number analyzed (Participants) | 742 | 765 | 764 | 743 | 743 | 764 | 746 | 761 | 731 | 776 | 706 | 801 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
score on a scale | 2.88 (0.05) | 2.73 (0.05) | 2.78 (0.05) | 2.70 (0.05) | 2.65 (0.05) | 2.68 (0.05) | 2.68 (0.05) | 2.68 (0.05) | 2.68 (0.06) | 2.74 (0.04) | 2.73 (0.05) | 2.74 (0.04) |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |

ADVERSE EVENTS:
Time Frame: From the time of consent up to about 4 weeks
Description: Participants will be randomized to see 6 packages and 10 advertisements with/without the claim of interest on each (32 arms). The randomization was repeated prior to each claim of interest. 1507 unique were enrolled in total. AEs are represented in male/female groups because it does not repeat as the arms do.
Groups:
- Male: Male participants
- Female: Female Participants
Arm/Group | Male | Female
All-Cause Mortality (participants affected / at risk) | 0/538 | 0/969
Serious Adverse Events (participants affected / at risk) | 0/538 | 0/969
Other Adverse Events (participants affected / at risk) | 0/538 | 0/969

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-16): https://cdn.clinicaltrials.gov/large-docs/21/NCT05439421/Prot_SAP_000.pdf